CLINICAL TRIAL: NCT06662500
Title: Prospective, Multicenter, Single-Arm, Investigational Device Exemption (IDE) Study of the Shockwave Intravascular Lithotripsy (IVL) System With the Shockwave Javelin Coronary IVL Catheter (FORWARD CAD IDE Study)
Brief Title: FORWARD CAD IDE Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 71886
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Intravascular Lithotripsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Shockwave Javelin Coronary IVL Catheter (Experimental): The Shockwave Javelin Coronary IVL Catheter will be used to treat subjects with moderate-to-severely calcified, stenotic de novo coronary artery lesions presenting with stable angina or following stabilization after acute coronary syndrome (ACS) that are suitable for non-emergent percutaneous coronary intervention (PCI).
  Interventions: Device: Intravascular Lithotripsy

INTERVENTIONS:
Device: Intravascular Lithotripsy — The Shockwave Intravascular Lithotripsy (IVL) System with the Shockwave Javelin Coronary Catheter is intended to treat calcified stenosis, including calcified stenoses that are anticipated to exhibit resistance to balloon crossing, full dilatation or subsequent uniform coronary stent expansion.

SUMMARY:
The FORWARD CAD IDE Study is a Prospective, Multicenter, Single-Arm, Investigational Device Exemption (IDE) Study conducted to assess the safety and effectiveness of the Shockwave Intravascular Lithotripsy (IVL) System with the Javelin Coronary IVL Catheter for the treatment of calcified, stenotic de novo coronary artery lesions prior to stenting.

DETAILED DESCRIPTION:
The Shockwave Javelin Coronary IVL Catheter was developed to address the current challenges clinicians face when treating tight, difficult to cross, calcified coronary lesions and was designed as a rapid exchange catheter to deliver intravascular lithotripsy to those complex lesions in the coronary vasculature.

The intended benefit of the Shockwave Javelin Coronary IVL Catheter is to allow the catheter to modify calcium in tight, difficult to cross lesions to increase the compliance of the vessel and allow further crossing of the device or additional treatment at the discretion of the physician.

Up to 158 subjects (150 evaluable) subjects with moderate-to severely calcified, stenotic de novo coronary artery lesions presenting with stable angina or following stabilization after acute coronary syndrome (ACS) that are suitable for non-emergent percutaneous coronary intervention (PCI) will be enrolled at up to 35 sites.

Once the pivotal cohort is fully enrolled (N=158), the study will continue to enroll an Extended Investigation cohort of up to 250 additional subjects.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subject is able and willing to comply with all assessments in the study.
3. Subjects with native coronary artery disease including stable angina or following stabilization after acute coronary syndromes (ACS) for non-emergent percutaneous coronary intervention (PCI)
4. Biomarkers (troponin) must be:

   1. less than or equal to the upper limit of lab normal within 24 hours prior to the procedure or may be drawn from the side port of the sheath at the time of index if the PCI is a non-emergent procedure and has stable angina (result will not be known prior to procedure); OR
   2. if above the upper limit of lab normal, biomarker result must be less than 5 times the upper limit of lab normal within 24 hours prior to the procedure and the following criteria must be met: • The procedure must not be emergent and the subject cannot have angina at rest.
5. Left ventricular ejection fraction (LVEF) >30% within 6 months (note: in the case of an event (MI or Revascularization) the LVEF must be taken post-event and in the case of multiple assessments of LVEF, the measurement closest to enrollment will be used for this criterion; may be assessed at time of index procedure).
6. Subject, or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures.
7. Estimated life expectancy >1 year.
8. Lesions in non-target vessels requiring PCI may be treated either:

   1. >30 days prior to the study procedure if the procedure was unsuccessful or complicated; OR
   2. >24 hours prior to the study procedure if the procedure was successful and uncomplicated (defined as a final lesion angiographic diameter stenosis <30% and TIMI 3 flow (visually assessed) for all non-target lesions and vessels without perforation, cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation, and no evidence of elevated biomarkers post-procedure; OR
   3. >30 days after the study procedure

   Angiographic Inclusion Criteria
9. The target lesion must be a de novo coronary lesion that has not been previously treated successfully with any interventional procedure
10. Single de novo target lesion stenosis of protected LMCA, or LAD, RCA or LCX (or of their branches)
11. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm
12. The target lesion must meet one of the following criteria:

    1. Target lesion stenosis >90% up to 40 mm in length and evidence of moderate or severe calcification at the lesion site. Moderate calcification defined as angiography with densities noted only during the cardiac cycle prior to contrast injection; severe calcification defined as angiography with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall; OR
    2. Chronic total occlusion presenting with J-CTO score of 1 with evidence of calcification and occlusion length up to 20 mm.
13. Guidewire must be in true lumen, distal to the lesion, and not subintimal, prior to insertion of Shockwave Javelin Coronary IVL catheter (antegrade wire technique only)

General Exclusion Criteria:

1. Any comorbidity or condition which may prevent compliance with this protocol, including follow-up visits
2. Subject is participating in another research study involving an investigational agent including pharmaceutical, biologic, or medical device that has not reached the primary endpoint
3. Subject is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment)
4. Unable to tolerate antiplatelet/anticoagulation therapy per society guidelines
5. Subject has an allergy to imaging contrast media which cannot be adequately pre-medicated
6. Subject experienced an acute STEMI within 30 days prior to index procedure
7. New York Heart Association (NYHA) class III or IV heart failure
8. Subject has acute or chronic renal disease with eGFR <30 ml/min/1.73m2 (using institutional formula)
9. History of a stroke or transient ischemic attack (TIA) within 60 days, or any prior intracranial hemorrhage or permanent neurologic deficit
10. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 3 months
11. Untreated pre-procedural hemoglobin <10 g/dL or intention to refuse blood transfusions if one should become necessary
12. Coagulopathy, including but not limited to platelet count <100,000 or International Normalized ratio (INR) >1.7 (INR is only required in subjects who have taken warfarin within 2 weeks of enrollment)
13. Subject has a hypercoagulable disorder such as polycythemia vera, platelet count >750,000 or other disorders
14. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics
15. Subjects with clinical evidence of cardiogenic shock
16. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
17. Subjects with an estimated life expectancy of less than 1 year
18. Non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days prior to the index procedure
19. Planned non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days after the index procedure
20. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
21. Planned use of atherectomy, scoring or cutting balloon, sub-intimal reentry device, or any investigational device other than coronary IVL

    Angiographic Exclusion Criteria
22. Unprotected left main diameter stenosis >30%
23. Evidence of a serious angiographic complication in the target vessel prior to treatment with coronary IVL (dissection, perforation, abrupt closure, persistent slow-flow or persistent no reflow)
24. Definite or possible thrombus by angiography in the target vessel
25. Evidence of aneurysm in target vessel within 10 mm of the target lesion
26. Second lesion with >50% stenosis in the same target vessel as the target lesion including its side branches
27. Chronic total occlusion of the target lesion, J-CTO ≥2
28. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
29. Previous stent within 5 mm of the target lesion
30. Failure to successfully cross the guidewire across the target lesion
31. Planned use of antegrade dissection and reentry (ADR), retrograde guidewire (RW), or retrograde dissection and reentry (RDR) crossing technique at any time during the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Freedom from MACE within 30 days | 30 Days
  Freedom from major adverse cardiac events (MACE) within 30 days of the index procedure. MACE (Clinical Events Committee [CEC] adjudicated) is defined as:
  * Cardiac death; or
  * Myocardial infarction (MI) defined as CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave at discharge (periprocedural MI) and using the Fourth Universal Definition of Myocardial Infarction beyond discharge (spontaneous MI); or
  * Target vessel revascularization (TVR) defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure
Primary Performance Endpoint - Technical Success | Peri-procedural
  Technical Success defined as successful Shockwave Javelin Coronary IVL-enabled lesion crossing without serious angiographic complications determined by angiographic core lab

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Yeh, M.D., M.Sc, M.B.A, Principal Investigator — Beth Israel Deaconess Medical Center; James C Spratt, MD, MB, ChB, FRCP, FESC, FACC, Principal Investigator — St. George's University NHS Trust; Robert F Riley, MD, MS, FACC, FAHA, FSCAI, Principal Investigator — Overlake Medical Center & Clinics
Locations (34):
- United States (28):
  - Scripps Health, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - South Denver Cardiology Associates, P.C, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital & Heart Center, Roslyn, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Providence St. Vincent, Portland, Oregon
  - Wellspan York Hospital, York, Pennsylvania
  - Centennial Heart, Nashville, Tennessee
  - Baylor Scott & White Research Institute Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott and White - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center Heart Institute, Salt Lake City, Utah
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Medical, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- United Kingdom (6):
  - Basildon University Hospital, Basildon, UK
  - Bristol Heart Institute, Bristol, UK
  - Leeds Teaching Hospital NHS Trust, Leeds, UK
  - Glenfield Hospital, Leicester, UK
  - St. Thomas Hospital, London, UK
  - St. George's Hospital, London, UK